CLINICAL TRIAL: NCT05298813
Title: A Randomized, Double-blind, Placebo-Controlled, Escalating Single Dose, Phase 1/2 Study to Evaluate the Efficacy and Safety of Inhaled IBIO123 in Participants With Mild to Moderate COVID-19 Illness
Brief Title: Phase 1/2 Study to Evaluate the Efficacy and Safety of Inhaled IBIO123 in Participants With Mild to Moderate COVID-19 Illness
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immune Biosolutions Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IBIO-INH-001
Record Dates: First submitted 2022-03-23; First posted 2022-03-28 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
Keywords: IBIO; IBIO123; mild COVID-19; moderate COVID-19; monoclonal antibodies; inhalation
MeSH Terms: conditions — COVID-19; Respiratory Aspiration | interventions — IBIO123

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental)
  Interventions: Biological: IBIO123
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: IBIO123 — IBIO123 1 mg, 5 mg and 10 mg
  Arms: Active
Other: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1/2, randomized, double-blind, placebo-controlled, single-dose escalating-dose study in participants with mild to moderate COVID-19 illness.

DETAILED DESCRIPTION:
Participants will be randomized to placebo or IBIO123.

In the phase 1 portion of the study, a total of 24 patients will be enrolled in 3 cohorts of 8 patients each. Six (6) of the 8 patients in each cohort will receive IBIO123 and 2 patients will receive placebo. The first cohort will be dosed with 1 mg. Subsequent cohorts will receive 5 mg, and 10 mg of IBIO123 or matching placebo and will be dosed at least 1 week apart to allow for review of safety and tolerability data for each prior cohort.

In the phase 2 portion of the study, as dose levels in phase 1 are determined to be safe, these dose levels may be introduced in phase 2 of Study IBIO-INH-001. This table describes the planned treatment arms. The Phase 2 portion of the study will enroll a total of approximately 200 participants (150 participants on study drug & 50 participants on Placebo).

ELIGIBILITY:
Inclusion Criteria:

Age

1. Are ≥18 years of age at the time of randomization

   Disease Characteristics
2. Are currently not hospitalized
3. Have one or more mild or moderate COVID-19 symptoms:

   i. Fever ii. Cough iii. Sore throat iv. Malaise v. Headache vi. Muscle pain vii. Gastrointestinal symptoms, or viii. Shortness of breath with exertion
4. Must have sample collection for first positive SARS-CoV-2 viral infection determination

   ≤3 days prior to start of the inhalation.

   Sex
5. Are men or non-pregnant women Reproductive and Contraceptive agreements and guidance is provided in Section 10.4, Appendix 4. Contraceptive use by men or women should be consistent with local regulations for those participating in clinical studies.

   Study Procedures
6. Understand and agree to comply with planned study procedures
7. Agree to the collection of nasopharyngeal swabs and venous blood Informed Consent
8. The participant or legally authorized representative gives signed informed consent as described in Section 14.1.3 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

   Exclusion Criteria:

   Medical Conditions
9. Have SpO2 ≤ 93% on room air, respiratory rate ≥30 per minute, resting heart rate ≥125 per minute.
10. Require mechanical ventilation or anticipated impending need for mechanical ventilation
11. Have known allergies to any of the components used in the formulation of the interventions.
12. Have hemodynamic instability requiring use of pressors within 24 hours of randomization.
13. Suspected or proven serious, active bacterial, fungal, viral, or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking intervention.
14. Have any co-morbidity requiring surgery or that is considered life- threatening within 29 days prior to dosing.
15. Have any serious concomitant systemic disease, condition or disorder that, in the opinion of the investigator, should preclude participation in this study.

    Other Exclusions
16. Have a history of a positive SARS-CoV-2 test prior to the one serving as eligibility for this study.
17. Have received an investigational intervention for SARS-CoV-2 prophylaxis within 30 days before dosing.
18. Have received treatment with a SARS-CoV-2 specific monoclonal antibody.
19. Have participated, within the last 30 days, in a clinical study involving an investigational intervention. If the previous investigational intervention has a long half-life, 5 half-lives or 30 days, whichever is longer, should have passed.
20. Are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
21. Are pregnant or breast feeding.
22. Are investigator site personnel directly affiliated with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Phase 1 : Characterize the effect of IBIO123 compared to placebo on safety and tolerability | From Baseline to Day 29
  Safety assessments such as AEs and SAEs
Phase 2: Characterize the effect of IBIO123 compared to placebo on SARS-CoV-2 viral load and viral clearance | From Baseline to Day 7
  Change from baseline to Day 7 in SARS-CoV-2 viral load

SECONDARY OUTCOMES:
Characterize the effect of IBIO123 compared to placebo on overall participant clinical status | From Baseline to Day 29
  Proportion (percentage) of participants who experience these events by Day 29:
  * COVID-19 related hospitalization (defined as ≥24 hours of acute care)
  * a COVID-19 related emergency room visit, or death
Characterize the effect of IBIO123 compared to placebo on SARS-CoV-2 viral load among participants with ≤8 days since symptom onset | From Baseline to Day 7
  Change from baseline to Day 7 in SARS-CoV-2 viral load among participants enrolled with ≤ 8 days of symptoms prior to randomization
Characterize the effect of IBIO123 compared to placebo on Baseline SARS-CoV-2 related symptoms | From Baseline to Day 29
  • Time to symptom reduction or resolution and proportion of patients
Characterize the effect of IBIO123 compared to placebo on SARS-CoV-2 viral load and viral clearance | From Baseline to Day 29
  • Proportion of participants who achieve SARS-CoV-2 clearance
Characterize the pharmacokinetics of IBIO123 | Days 1, 3, 7, and 29
  IBIO123 mean plasma concentration
Phase 1: Characterize the effect of IBIO123 compared to placebo on SARS-CoV-2 viral load and viral clearance | From Baseline to Day 7
  Change from baseline to Day 7 in SARS-CoV-2 viral load
Phase 2 : Characterize the effect of IBIO123 compared to placebo on safety and tolerability | From Baseline to Day 29
  Safety assessments such as AEs and SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Labbe, PhD, Study Director — Immune Biosolutions
Locations (11):
- Brazil (5):
  - Santa Casa de Misercórdia de Passos, Passos, Minas Gerais
  - Instituto Brasil de Pesquisa Clinica, Glória, Rio de Janeiro
  - Clinica Supera Oncologia, Chapecó, Santa Catarina
  - Instituto Brasileiro de Controle do Câncer / Sao Camilo Oncologia, Pompéia, São Paulo
  - Pesquisare Saúde, Santo André, São Paulo
- South Africa (6):
  - FARMOVS, Bloemfontein, Free State
  - Newton Clinical Trial Centre, Newtown, Gauteng
  - Johese Clinical Research ZAH, Pretoria, Gauteng
  - Jongaie Research, Pretoria West, Gauteng
  - Durban International Clinical Research, Enhancing Care Foundation, Durban, KwaZulu-Natal
  - Clinical Research Institute of South Africa - CRISA, KwaDukuza, KwaZulu-Natal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maranda B, Labbe SM, Lurquin M, Brabant P, Fugere A, Larrivee JF, Grbic D, Leroux A, Leduc F, Finzi A, Gaudreau S, Swart Y; IBIO-INH-001 Investigators. Safety and efficacy of inhaled IBIO123 for mild-to-moderate COVID-19: a randomised, double-blind, dose-ascending, placebo-controlled, phase 1/2 trial. Lancet Infect Dis. 2024 Jan;24(1):25-35. doi: 10.1016/S1473-3099(23)00393-6. Epub 2023 Aug 21. PMID 37619584